CLINICAL TRIAL: NCT07327918
Title: Effect of Epidural Needle Injection on Catheter Placement Success During Painless Labour: A Prospective Randomized Study
Brief Title: Effect of Epidural Needle Injection on Catheter Placement Success During Painless Labour
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC.11.9.2025
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Labour Analgesia
Keywords: Epidural Needle
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection group (Experimental): Patients will receive [10 ml of local anaesthetic] through an epidural needle before catheter advancement.
  Interventions: Procedure: Injection Group
- Control group (Placebo Comparator): No injection before catheter insertion.
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Injection Group — Patients will receive [10 ml of local anesthetic] through an epidural needle before catheter advancement.
  Arms: Injection group
Other: Control group — No injection before catheter insertion.
  Arms: Control group

SUMMARY:
Epidural analgesia is the gold standard for painless labour, but successful catheter placement can be technically challenging due to anatomical and physiological changes in pregnancy. Injecting saline or local anesthetic through the epidural needle before catheter insertion has been proposed to facilitate catheter advancement by dilating the epidural space. This study aimed to evaluate the effect of epidural needle injection on the success rate and ease of catheter placement during labour analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-40 years.
* ASA physical status II or III.
* Singleton pregnancy.
* Gestational age ≥37 weeks.
* Active labour with cervical dilatation ≥3 cm.
* Cephalic presentation.
* Requesting epidural analgesia for painless labour.
* Ability to provide written informed consent.

Exclusion Criteria:

* • Refusal to participate or to sign informed consent.

  * Age <18 or >40 years.
  * ASA status ≥IV.
  * Allergy to local anesthetics or saline.
  * Coagulopathy or platelet count <100,000/mm³.
  * Local infection at the insertion site.
  * Severe spinal deformity (scoliosis, kyphosis).
  * Multiple pregnancy.
  * Non-cephalic presentation (breech, transverse).
  * Antepartum hemorrhage or placenta previa.
  * Severe preeclampsia or eclampsia.
  * Signs of fetal distress.
  * Previous lumbar spine surgery.
  * Difficult epidural anatomy (on ultrasound or palpation).
  * BMI >40 kg/m²

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Painless Labour
Enrollment: 216 (Estimated)
Dates: Start 2026-06-28 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Success of epidural catheterization on the first attempt. | Assessed immediately during the procedure at the time of epidural catheter placement.
  The incidence of success of epidural catheterization on the first attempt will be determined. This measures whether the epidural catheter is successfully inserted on the first attempt after loss of resistance, without the need for repositioning or reattempt. Success is defined by obtaining adequate analgesia with proper catheter function (confirmed by clinical effect).

SECONDARY OUTCOMES:
Number of catheterization attempts | Assessed during the procedure until successful catheterization is achieved.
  Counts the total number of insertion attempts required to achieve correct epidural catheter placement, reflecting technical ease and procedural efficiency.
Procedure duration | Assessed intraoperatively, recorded from the beginning of the puncture until catheter fixation.
  Measures the time elapsed between needle insertion and successful catheter placement, expressed in minutes. Shorter duration indicates greater ease of insertion.
Incidence of numbness | Assessed post-catheter insertion, within the first 30 minutes after drug administration.
  Records any occurrence of unexpected or abnormal sensory numbness following the epidural test dose or analgesic administration, which may indicate uneven drug spread or misplaced catheter.
Incidence of unintended dural puncture | Assessed immediately at the time of needle insertion or catheter placement.
  Identifies accidental dural puncture events occurring during epidural space entry or catheter advancement.
Maternal satisfaction | Assessed post-delivery, usually within 24 hours after labour.
  Evaluates the mother's satisfaction regarding the analgesia quality, comfort during the procedure, and overall experience. Typically rated using a structured satisfaction scale. Maternal satisfaction can be measured on a 0-5 scale using a simple 5-point Likert-type item: 0 = completely dissatisfied, 1 = dissatisfied, 2 = neutral, 3 = satisfied, and 4 = very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP